CLINICAL TRIAL: NCT02459353
Title: Effect of Dapagliflozin on Glycemic Variability as an add-on Therapy in Subjects With Type 2 Diabetes Mellitus With in Inadequate Glycemic Control in Insulin: a Multicenter, Placebo-controlled, Double-blind, Randomized Study
Brief Title: Effect of Dapagliflozin on Glycemic Variability
Acronym: DIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: AstraZeneca (Industry); Severance Hospital (Other); Eulji General Hospital (Other); Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Kun-Ho Yoon, Professor of endocrinology division, Department of Internal Medicine, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISSDAPA0006
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: dapagliflozin; glucose variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dapagliflozin 10mg (Experimental): a group which treated with dapagliflozin 10mg plus basal insulin therapy
  Interventions: Drug: Dapagliflozin
- placebo 10mg (Placebo Comparator): a group which treated with dapagliflozin placebo plus basal insulin therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin
  Arms: dapagliflozin 10mg
Drug: Placebo
  Arms: placebo 10mg

SUMMARY:
Dapagliflozin improves glycemic variability in subjects with type 2 diabetes mellitus when added to insulin therapy. The primary objective of this study is to assess the effect of dapagliflozin on glucose variability compared to placebo after 12 weeks of treatment in type 2 diabetic patients with inadequate glycemic control on insulin.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled phase 4 study to evaluate whether treatment with dapagliflozin add-on to insulin reduces glucose variability in type 2 Diabetes Mellitus. The study will recruit type 2 Diabetes Mellitus patients with inadequate glucose control on insulin treatment with or without metformin or sulphonylurea. It is estimated that 90 type 2 diabetic patients will be enrolled. After randomization, a total 12 week treatment of dapagliflozin or matching placebo will be administered. Before and after treatment, tests for efficacy and safety outcomes will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male aged 20~70 years
2. Type 2 diabetes patients
3. Treatment on basal insulin therapy ≥0.2U/kg/day(±metformin and/or ±sulfonylurea) for at least 12 weeks
4. Inadequate glycemic control ; HbA1c 7.0%~10.0% at screening
5. Female of childbearing potential agrees to routinely use of adequate contraception from signing of the informed consent throughout the duration of the study
6. Understands the study procedure, alternatives, and risks and voluntarily agrees to participated by giving written informed consent

Exclusion Criteria:

1. Type 1 diabetes(Fasting C-peptide ≤ 0.78ng/dL(or 0.26 nM/L)), secondary diabetes, gestational diabetes
2. Insulin therapy modalities containing short or rapid acting insulin (continuous subcutaneous insulin injection, pre-mixed insulin, basal-bolus insulin)
3. History of diabetic ketoacidosis, hyperglycemic hyperosmolar state
4. Estimated glomerular filtration rate <60 mL/min/1.73 m2
5. History of chronic cystitis or recurrent urinary tract infection
6. Currently on loop diuretics
7. Adrenal insufficiency, pituitary insufficiency
8. Currently on medication known to affect glucose metabolism (e.g. corticosteroids, immunosuppressants)
9. Hemoglobin <10g/dL in female, <12g/dL in male
10. Abnormal liver function (AST/ALT > x3 upper normal limit)
11. On weight loss program or taking weight loss medication
12. NYHA class III, IV congestive heart failure
13. History of acute myocardial infarction, unstable angina, coronary artery bypass graft or stroke within 6 months
14. History of bladder cancer
15. History of malignancy within 5 years
16. Pregnant or lactating women
17. History of excessive alcohol abuse (≥30g/day)
18. Hypersensitivity to SGLT2 inhibitors
19. Patient with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
20. Subject who the investigator deems inappropriate to participate in this study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Glycemic Variability (mean amplitude of glycemic excursion) | baseline and 12 weeks
  MAGE(mean amplitude of glycemic excursion)
Glycemic Variability (Coefficient of Variation) | baseline and 12 weeks
  CV (Coefficient of Variation)
Glycemic Variability (Standard Deviation) | baseline and 12 weeks
  SD (Standard Deviation)

SECONDARY OUTCOMES:
glycemic control variables HbA1C | baseline and each visit(6weeks, 12weeks)
  HbA1C
glycemic control variables Fasting Plasma Glucose | baseline and each visit(6weeks, 12weeks)
  Fasting Plasma Glucose
lipid profile Total cholesterol | baseline and each visit(6weeks, 12weeks)
  Total cholesterol
lipid profile Triglyceride | baseline and each visit(6weeks, 12weeks)
  Triglyceride
lipid profile HDL-cholesterol | baseline and each visit(6weeks, 12weeks)
  HDL-cholesterol
lipid profile LDL-cholesterol | baseline and each visit(6weeks, 12weeks)
  LDL-cholesterol
glycemic control variables Percentage of patients achieving HbA1c < 7% | 12weeks
  Percentage of patients achieving HbA1c < 7%
glycemic control variables Percentage of patients achieving HbA1c < 6.5% | 12weeks
  Percentage of patients achieving HbA1c < 6.5%
glycemic control variables 24hr urinary glucose excretion | baseline and 12weeks
  24hr urinary glucose excretion
glycemic control variables Changes in insulin dose | baseline and each visit(6weeks, 12weeks)
  Changes in insulin dose
blood pressure SBP | baseline and each visit(6weeks, 12weeks)
  SBP
blood pressure DBP | baseline and each visit(6weeks, 12weeks)
  DBP

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ho Yoon, Ph.D., Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seoul, South Korea